CLINICAL TRIAL: NCT04313855
Title: Help With Early Detection of Postoperative Neuropathic Pain Using SMS After Ambulatory Surgery
Acronym: SMS DPpostop
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SMS DPpostop
Record Dates: First submitted 2020-03-16; First posted 2020-03-18 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Chronic Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: This is a prospective case-control diagnostic study nestled in a cohort. The cohort is the set of patients operated on ambulatory surgery on the GHPSJ. In this cohort, pain patients according to the doctor's opinion are the cases. The controls are the patients who are not painful according to the doctor's opinion.
  For reasons of available consultation time slots, it is not possible to see all of the patients. It was therefore decided to see all the painful patients and to select by lot the painless patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chronic post-operative pain (Experimental): 7 days after the intervention, the patient receives a standardized questionnaire by SMS, to determine whether the patient has pain at the operating site and whether this pain has the characteristics of neuropathic pain. After replying to the SMS, the patient will be contacted by phone to assess: the intensity of pain at the operating site using a numerical scale and the existence of neuropathic pain. Depending on the responses received by SMS and/or phone, a consultation appointment with an anesthesiologist specializing in pain may be offered within a maximum of 2 weeks.
  Ninety days after your surgery, the patient receives the same standardized questionnaire by SMS. The patient will be contacted by telephone, in order to assess the intensity of pain at the operating site and the existence of neuropathic pain using. If the patient has post-operative pain, a consultation appointment with an anesthesiologist specializing in pain will be offered to him within a maximum of 2 weeks.
  Interventions: Diagnostic Test: SMS in the early detection of postoperative neuropathic pain

INTERVENTIONS:
Diagnostic Test: SMS in the early detection of postoperative neuropathic pain — 7 days after the intervention, the patient receives a standardized questionnaire by SMS, to determine whether the patient has pain at the operating site and whether this pain has the characteristics of neuropathic pain. After replying to the SMS, the patient will be contacted by phone to assess: the intensity of pain at the operating site using a numerical scale and the existence of neuropathic pain. Depending on the responses received by SMS and/or phone, a consultation appointment with an anesthesiologist specializing in pain may be offered within a maximum of 2 weeks.
  Ninety days after your surgery, the patient receives the same standardized questionnaire by SMS. The patient will be contacted by telephone, in order to assess the intensity of pain at the operating site and the existence of neuropathic pain using. If the patient has post-operative pain, a consultation appointment with an anesthesiologist specializing in pain will be offered to him within a maximum of 2 weeks.

SUMMARY:
Chronic post-operative pain is generally defined by persistent pain more than 2 months after surgery. General reviews on chronic post-operative pain describe an overall incidence of 30%, of which 5 to 10% are described as severe. Different risk factors have been identified: pain and preoperative opioid use, anxiety - depression, catastrophism, type of surgery, intensity and duration of postoperative pain, genetic factors.

If postoperative pain is essentially pain caused by excess nociceptive stimulation, investigators realize that a neuropathic component is far from being exceptional and that this can be demonstrated quickly after surgery. In addition, these neuropathic pains respond little or no to the usual analgesics and in particular to opioids, which can be the cause of misuse or death from overdose. Early detection of pain of a neuropathic nature would allow appropriate therapy to be put in place and may therefore reduce the risk of chronic postoperative pain.

The concept of ambulatory surgery assumes that postoperative pain will be minimal and can be controlled at home by the administration of oral pain relievers. However, following the development of surgical techniques and the improvement in the quality of care, the number and complexity of procedures that can be performed in ambulatory surgery have increased considerably. Consequently, a significant number of patients will probably develop chronic post-operative pain without the possibility of early detection. The prevalence of chronic post-operative pain in ambulatory surgery has been studied by a single team. The authors conclude that it is underestimated and variable depending on the surgery between 15 and 32%.

For the past few years, the GHPSJ has been using an ambulatory surgery algorithm that sends SMS messages to warn and follow up on patients. The principle is simple: patients scheduled for outpatient surgery receive text messages the day before their intervention to remind them of the instructions to be followed and the meeting times and, the day after the operation, the algorithm sends SMS to ask patients if all is well or if they have pain, nausea or vomiting, discharge from the scar. In postoperative monitoring, this technology has shown promising results.

This technology has not been used in the screening of persistent pain. The objective of this work is to assess the effectiveness of an SMS algorithm in the early detection of postoperative neuropathic pain after surgery performed on an outpatient basis.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged ≥ 18 years
* Patient hospitalized on an outpatient basis within the Paris Saint Joseph Hospital Group in the following different surgical specialties: orthopedics, digestive, vascular, gynecological, plastic and restorative
* French speaking patient
* Patient with smartphone
* Patient affiliated to a social security scheme
* Patient having given oral, free, informed and express consent

Exclusion Criteria:

* Patient under guardianship or curatorship
* Patient deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Actual)
Dates: Start 2020-12-09 (Actual); Primary Completion 2022-07-07 (Actual); Study Completion 2022-10-28 (Actual)

PRIMARY OUTCOMES:
diagnostic method | Day 7
  This outcome corresponds to the calculation of the sensitivity and the specificity of the diagnostic method tested which is the combination of SMS and the DN2 questionnaire.

SECONDARY OUTCOMES:
Persistent post-surgical pain day 90 | Day 90
  This oucome correspond to corresponds to the proportion of patients with persistent post-surgical pain at seven days after surgery performed on an outpatient basis.
Neuropathic pain day90 | Day 90
  This outcome correspond to the proportion of neuropathic pain on Day90 estimated using the questionnaires DN4 and NPSI during the postoperative pain consultation.
signs suggestive of neuropathic pain day90 | Day 90
  This outcome correspond to the proportion of patients with signs suggestive of neuropathic pain during the consultation carried out by an anesthesiologist specialized in pain 90 days after the intervention.
Comparison of pain between day7 and day90 | Day90
  This outcome corresponds to the comparison of the proportion of patients with signs suggestive of neuropathic pain during the consultation carried out by an anesthesiologist specialized in pain between Day7 and Day90 after the intervention.
Proportion of patients presenting signs suggestive of pain | Day90
  This ouctome corresponds to the proportion of patients presenting signs suggestive of neuropathic pain during the consultation carried out by an anesthesiologist specialized in pain on Day90 who had presented pain on Day7.

CONTACTS AND LOCATIONS:
Overall Officials: Frederic ADAM, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, France

REFERENCES:
- [Result] Macrae WA. Chronic post-surgical pain: 10 years on. Br J Anaesth. 2008 Jul;101(1):77-86. doi: 10.1093/bja/aen099. Epub 2008 Apr 22. PMID 18434337
- [Result] Johansen A, Romundstad L, Nielsen CS, Schirmer H, Stubhaug A. Persistent postsurgical pain in a general population: prevalence and predictors in the Tromso study. Pain. 2012 Jul;153(7):1390-1396. doi: 10.1016/j.pain.2012.02.018. Epub 2012 Mar 24. PMID 22445291
- [Result] Fletcher D, Stamer UM, Pogatzki-Zahn E, Zaslansky R, Tanase NV, Perruchoud C, Kranke P, Komann M, Lehman T, Meissner W; euCPSP group for the Clinical Trial Network group of the European Society of Anaesthesiology. Chronic postsurgical pain in Europe: An observational study. Eur J Anaesthesiol. 2015 Oct;32(10):725-34. doi: 10.1097/EJA.0000000000000319. PMID 26241763
- [Result] Glare P, Aubrey KR, Myles PS. Transition from acute to chronic pain after surgery. Lancet. 2019 Apr 13;393(10180):1537-1546. doi: 10.1016/S0140-6736(19)30352-6. PMID 30983589
- [Result] Beloeil H, Sion B, Rousseau C, Albaladejo P, Raux M, Aubrun F, Martinez V; SFAR research network. Early postoperative neuropathic pain assessed by the DN4 score predicts an increased risk of persistent postsurgical neuropathic pain. Eur J Anaesthesiol. 2017 Oct;34(10):652-657. doi: 10.1097/EJA.0000000000000634. PMID 28437260
- [Result] Hoofwijk DM, Fiddelers AA, Peters ML, Stessel B, Kessels AG, Joosten EA, Gramke HF, Marcus MA. Prevalence and Predictive Factors of Chronic Postsurgical Pain and Poor Global Recovery 1 Year After Outpatient Surgery. Clin J Pain. 2015 Dec;31(12):1017-25. doi: 10.1097/AJP.0000000000000207. PMID 25565589
- [Result] Hoofwijk DMN, Fiddelers AAA, Emans PJ, Joosten EA, Gramke HF, Marcus MAE, Buhre WFFA. Prevalence and Predictive Factors of Chronic Postsurgical Pain and Global Surgical Recovery 1 Year After Outpatient Knee Arthroscopy: A Prospective Cohort Study. Medicine (Baltimore). 2015 Nov;94(45):e2017. doi: 10.1097/MD.0000000000002017. PMID 26559300
- [Result] Lu K, Marino NE, Russell D, Singareddy A, Zhang D, Hardi A, Kaar S, Puri V. Use of Short Message Service and Smartphone Applications in the Management of Surgical Patients: A Systematic Review. Telemed J E Health. 2018 Jun;24(6):406-414. doi: 10.1089/tmj.2017.0123. Epub 2017 Nov 7. PMID 29111887
- [Result] Carrier G, Cotte E, Beyer-Berjot L, Faucheron JL, Joris J, Slim K; Groupe Francophone de Rehabilitation Amelioree apres Chirurgie (GRACE). Post-discharge follow-up using text messaging within an enhanced recovery program after colorectal surgery. J Visc Surg. 2016 Aug;153(4):249-52. doi: 10.1016/j.jviscsurg.2016.05.016. Epub 2016 Aug 8. PMID 27423211
- [Result] Chen Y, Chin M, Greenberg S, Johnstone C, McGuinness J. Post-tonsillectomy pain in 24 children - utilising short message service (SMS) to assess postoperative outcomes. Clin Otolaryngol. 2012 Oct;37(5):412-4. doi: 10.1111/j.1749-4486.2012.02521.x. No abstract available. PMID 23164270
- [Result] Bouhassira D, Attal N, Alchaar H, Boureau F, Brochet B, Bruxelle J, Cunin G, Fermanian J, Ginies P, Grun-Overdyking A, Jafari-Schluep H, Lanteri-Minet M, Laurent B, Mick G, Serrie A, Valade D, Vicaut E. Comparison of pain syndromes associated with nervous or somatic lesions and development of a new neuropathic pain diagnostic questionnaire (DN4). Pain. 2005 Mar;114(1-2):29-36. doi: 10.1016/j.pain.2004.12.010. Epub 2005 Jan 26. PMID 15733628
- [Result] Wall PD, Sprowson AP, Parsons N, Parsons H, Achten J, Balasubramanian S, Costa ML; Perioperative Analgesia for Knee Arthroplasty Collaborators. Protocol for a single-centre randomised controlled trial of multimodal periarticular anaesthetic infiltration versus single-agent femoral nerve blockade as analgesia for total knee arthroplasty: Perioperative Analgesia for Knee Arthroplasty (PAKA). BMJ Open. 2015 Dec 21;5(12):e009898. doi: 10.1136/bmjopen-2015-009898. PMID 26692559
- [Result] Remerand F, Godfroid HB, Brilhault J, Vourc'h R, Druon J, Laffon M, Fusciardi J. Chronic pain 1 year after foot surgery: Epidemiology and associated factors. Orthop Traumatol Surg Res. 2014 Nov;100(7):767-73. doi: 10.1016/j.otsr.2014.07.012. Epub 2014 Oct 8. PMID 25306303
- [Result] van Zaane B, Vergouwe Y, Donders AR, Moons KG. Comparison of approaches to estimate confidence intervals of post-test probabilities of diagnostic test results in a nested case-control study. BMC Med Res Methodol. 2012 Oct 31;12:166. doi: 10.1186/1471-2288-12-166. PMID 23114025